CLINICAL TRIAL: NCT04680923
Title: Efficacy of Combined Periportal and Preperitoneal Local Anesthetic Infiltration (CPPLAI) in Laparoscopic Sleeve Gastrectomy Patients
Brief Title: Efficacy of CPPLAI in Laparoscopic Sleeve Gastrectomy Patients
Acronym: CPPLAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khalid University Hospital (Other)
Responsible Party: Principal Investigator, Abdul Sattar Narejo, Consultant Anesthesiologist, King Khalid University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Project No. E-20-5332
Record Dates: First submitted 2020-12-08; First posted 2020-12-23 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Obesity, Morbid; Pain, Postoperative
Keywords: Laparoscopic sleeve gastrectomy; post operative pain; local anesthetic infiltration; Periportal; Preperitoneal; Morbid obesity
MeSH Terms: conditions — Obesity, Morbid; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: 117 adult patients scheduled for Laparoscopic Sleeve Gastrectomy (LSG) will be recruited in this prospective clinical study. The patients will be divided into two groups; group-1 (CPPLAI) (n= 59) will receive intraoperative combined periportal and preperitoneal bupivacaine 0.25% 2-3 mg/kg diluted in 40 ml normal saline and group 2 (placebo) (n= 58) periportal and preperitoneal 40 ml of sterile water will be injected.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All patients, care providers in PACU & ward (nurses), and outcome assessors (assistant anesthesiologist) will be blinded to the group allocation. Only the assigned anesthesiologist responsible for perioperative care and the surgeon performing preperitoneal local anesthetic infiltration will be aware of the group allocation to treat any unwanted side effects during and after the operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPPLAI (Experimental): Group-1 (CPPLAI) (n= 59) will receive intraoperative combined periportal and preperitoneal bupivacaine 0.25% 2-3 mg/kg diluted in 40 ml normal saline in patients scheduled for laparoscopic sleeve gastrectomy.
  Interventions: Procedure: CPPLAI; Drug: Bupivacaine 0.25%
- Placebo (Placebo Comparator): Group 2 (placebo) (n= 58) will receive intraoperative combined periportal and preperitoneal sterile water 40 ml in patients scheduled for laparoscopic sleeve gastrectomy.
  Interventions: Other: Placebo

INTERVENTIONS:
Procedure: CPPLAI — In this intervention, after general anesthesia patients will receive intraoperative combined periportal and preperitoneal bupivacaine 0.25% 2-3 mg/kg diluted in 40 ml normal saline.
  Other Names: Bupivacaine 0.25%
  Arms: CPPLAI
Other: Placebo — In this intervention, after general anesthesia patients will receive intraoperative combined periportal and preperitoneal 40 ml of sterile water.
  Other Names: Sterile water
  Arms: Placebo
Drug: Bupivacaine 0.25% — In this intervention, after general anesthesia patients will receive intraoperative combined periportal and preperitoneal bupivacaine 0.25% 2-3 mg/kg diluted in 40 ml normal saline.
  Other Names: CPPLAI
  Arms: CPPLAI

SUMMARY:
The high demand for bariatric surgery due to the increasing prevalence of obesity worldwide necessitate evidence-based clinical pathway such as Enhanced Recovery After Bariatric Surgery (ERABS). The paradigm of surgery has been shifted from open to laparoscopic in morbidly obese patients. Laparoscopic Sleeve Gastrectomy (LSG) is the most common procedure performed in our institute for sustained weight loss and amelioration of obesity-related comorbidities. Pain control in ERABS is one of the key factors for improved outcomes. Surgery induced acute postoperative pain, stress response and fatigue lead to prolonged convalescence and hospital stay. Optimal titrated safe postoperative pain management in LSG patients still remains a challenge.

DETAILED DESCRIPTION:
Obesity is a complex multifactorial disease. The worldwide prevalence of obesity has doubled since 1980 to a level that now almost a third of the world's population is classified as overweight. Laparoscopic Sleeve Gastrectomy (LSG) is one of the effective treatments for sustained weight loss and to ameliorate the obesity-related comorbidities, and now the most commonly performed bariatric surgery worldwide. Postoperative pain from the laparoscopic portal sites and the visceral pain after gastrectomy requires a multimodal approach for pain management. As obese patients are sensitive to opioids overdose and at risk of respiratory depression and obstructive sleep apnoea, local anesthetic infiltration at the surgical incision sites and preperitoneal can decrease postoperative opioid consumption after LSG. Perioperative multimodal analgesia uses combinations of analgesic medications that act on different sites and pathways in an additive or synergistic manner to achieve pain relief with minimal or no opiate consumption. Although all medications have side effects, opiates have particularly concerning, multisystemic, long-term, and short-term side effects, which increase morbidity and prolong admissions. local infiltration analgesia (LIA) used widely as an effective component of multimodal analgesia and represents valuable options for controlling perioperative pain. LIA involves the injection and/or infusion of a local anesthetic near the site of surgical incision to provide targeted analgesia. A wide variety of techniques have been described, including single-injection intraoperative wound infiltration, indwelling wound infusion catheters, and the recent high-volume LIA technique associated with joint replacement surgery. Although, preperitoneal local anesthetic infiltration is a novel technique that was first described for pain relief after laparoscopic hernia repair. Recently, the investigators have used this technique in our institute during laparoscopic hernia repair which is now gaining popularity worldwide. Another investigator reported that continuous preperitoneal analgesia better attenuated postoperative inflammatory response and provided comparable overall analgesia to that with continuous epidural analgesia following radical cystectomy. Recently, a large systematic review and meta-analysis comparing preperitoneal or subcutaneous wound catheters with epidural analgesia in abdominal surgery showed preperitoneal wound catheters are an effective pain modality in abdominal surgery. Pain control was as effective as epidural analgesia and recovery parameters, opioid consumption, the incidence of hypotension, and patient satisfaction seemed to be in favor of preperitoneal wound catheters compared with active alternatives, as well as placebo. The trend for bariatric surgery is now moving towards opiates-almost free anesthesia. Since the first description of preperitoneal local anesthetic infiltration almost 2 decades ago little work has been done to test its efficacy, especially in LSG patients. The investigators of this study hypothesis that CPPLAI is an effective technique to reduce postoperative pain and favors early mobilization and patient satisfaction due to its fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status I-III
* Age 18-60 years
* Either gender
* Obese patients (BMI >35 for laparoscopic sleeve gastrectomy

Exclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status IV
* Patients uncontrolled HTN
* Anticipated difficult intubation
* Allergic to morphine
* Clinically significant neurological, cardiovascular, renal hepatic disease planned for postoperative surgical intensive care (SICU) admission
* History of drug abuse or chronic opioid use

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | From preoperative to day two postoperative
  Pain will be measured postoperatively using numerical rating scale (NRS) from 0 to 10 after laparoscopic sleeve gastrectomy. Where 0 is no pain and 10 is worst pain imaginable.

SECONDARY OUTCOMES:
Postoperative Morphine consumption | From preoperative to day two postoperative
  Postoperative intravenous Morphine consumption in milligrams will be calculated as a total dose per patient that received to control pain after laparoscopic sleeve gastrectomy.
Length of hospital stay | Through study completion, an average of 2 days.
  Total number of days the patient stay in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Sattar Narejo, FCPS, Principal Investigator — King Khalid University Hospital
Locations (1):
- King Khalid University Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
After completing the data collection by July 2021, Pain score, opioid consumption, and length of hospital stay will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: December 2021
Access Criteria: IPD (protocol, statistical analysis) will be shared on submitting requests through email to the principal investigator.

REFERENCES:
- [Background] Chooi YC, Ding C, Magkos F. The epidemiology of obesity. Metabolism. 2019 Mar;92:6-10. doi: 10.1016/j.metabol.2018.09.005. Epub 2018 Sep 22. PMID 30253139
- [Background] Chung AY, Thompson R, Overby DW, Duke MC, Farrell TM. Sleeve Gastrectomy: Surgical Tips. J Laparoendosc Adv Surg Tech A. 2018 Aug;28(8):930-937. doi: 10.1089/lap.2018.0392. Epub 2018 Jul 13. PMID 30004814
- [Background] Belcaid I, Eipe N. Perioperative Pain Management in Morbid Obesity. Drugs. 2019 Jul;79(11):1163-1175. doi: 10.1007/s40265-019-01156-3. PMID 31256367
- [Background] Boerboom SL, de Haes A, Vd Wetering L, Aarts EO, Janssen IMC, Geurts JW, Kamphuis ET. Preperitoneal Bupivacaine Infiltration Reduces Postoperative Opioid Consumption, Acute Pain, and Chronic Postsurgical Pain After Bariatric Surgery: a Randomized Controlled Trial. Obes Surg. 2018 Oct;28(10):3102-3110. doi: 10.1007/s11695-018-3341-6. PMID 29926357
- [Background] Beverly A, Kaye AD, Ljungqvist O, Urman RD. Essential Elements of Multimodal Analgesia in Enhanced Recovery After Surgery (ERAS) Guidelines. Anesthesiol Clin. 2017 Jun;35(2):e115-e143. doi: 10.1016/j.anclin.2017.01.018. PMID 28526156
- [Background] Merritt CK, Mariano ER, Kaye AD, Lissauer J, Mancuso K, Prabhakar A, Urman RD. Peripheral nerve catheters and local anesthetic infiltration in perioperative analgesia. Best Pract Res Clin Anaesthesiol. 2014 Mar;28(1):41-57. doi: 10.1016/j.bpa.2014.02.002. Epub 2014 Mar 18. PMID 24815966
- [Background] Joshi GP, Machi A. Surgical site infiltration: A neuroanatomical approach. Best Pract Res Clin Anaesthesiol. 2019 Sep;33(3):317-324. doi: 10.1016/j.bpa.2019.07.017. Epub 2019 Jul 25. PMID 31785717
- [Background] Deans GT, Wilson MS, Brough WA. Controlled trial of preperitoneal local anaesthetic for reducing pain following laparoscopic hernia repair. Br J Surg. 1998 Jul;85(7):1013-4. doi: 10.1046/j.1365-2168.1998.00763.x. PMID 9692587
- [Background] Aldohayan A, Eldawlatly A. Combined preincisional periportal and preperitoneal infiltration with bupivacaine in pain relief after laparoscopic surgery. Saudi J Anaesth. 2017 Apr-Jun;11(2):135-136. doi: 10.4103/sja.SJA_153_17. No abstract available. PMID 28442949
- [Background] Othman AH, Ahmed DG, Abd El-Rahman AM, El Sherif FA, Mansour S, Aboeleuon E. Effect of Preperitoneal Versus Epidural Analgesia on Postoperative Inflammatory Response and Pain Following Radical Cystectomy: A Prospective, Randomized Trial. Clin J Pain. 2019 Apr;35(4):328-334. doi: 10.1097/AJP.0000000000000679. PMID 30829734
- [Background] Mungroop TH, Bond MJ, Lirk P, Busch OR, Hollmann MW, Veelo DP, Besselink MG. Preperitoneal or Subcutaneous Wound Catheters as Alternative for Epidural Analgesia in Abdominal Surgery: A Systematic Review and Meta-analysis. Ann Surg. 2019 Feb;269(2):252-260. doi: 10.1097/SLA.0000000000002817. PMID 29781846
- [Background] Lirk P, Rathmell JP. Opioid-free anaesthesia: Con: it is too early to adopt opioid-free anaesthesia today. Eur J Anaesthesiol. 2019 Apr;36(4):250-254. doi: 10.1097/EJA.0000000000000965. No abstract available. PMID 30817360